CLINICAL TRIAL: NCT04060810
Title: Value of MRI CSF Flowmetry in Assessment of Grey Zone Hydrocephalic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Hossam Mohammad Hassan, Resident at neurosurgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: grey zone hydrocephalus
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus | interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- grey zone hydrocephalic patients (Other): MR CSF flowmetry CT brain Ventriculoperitoneal shunt
  Interventions: Other: MR CSF flowmetry

INTERVENTIONS:
Other: MR CSF flowmetry — MR flowmetry in grey zone hydro cephalic patients followed by ventriculoperitoneal shunt
  Other Names: CT brain; Ventriculoperitoneal shunt

SUMMARY:
To evaluate accuracy of (MRI) cerebrospinal fluid flowmetry after shunt operation in patients with borderline (grey zone) hydrocephalus.

DETAILED DESCRIPTION:
Hydrocephalus could be defined as disturbance of formation, flow or absorption of CSF. We encounter some challenging cases with intermittent non specific symptoms as delayed milestones and headache with concomitant imaging showing dilated ventricular system, so we find ourselves hesitating to take the decision of surgical intervention to put shunt or not, therefore MRI CSF flowmetry gives us a chance to overcome this problem. Phase contrast MR imaging is a rapid, simple and non-invasive technique which is sensitive to even small CSF flows, and can be used to evaluate CSF flow both qualitatively and quantitatively.

CSF flow measurement at the suspected level of obstruction gives reliable and reproducible results for more accurate diagnosis and can be used to guide therapeutic decisions in a more reliable manner, and follow up post treatment outcome.

With the CT and magnetic resonance imaging (MRI) techniques, it is possible to localize with accuracy the exact site of blockage of flow to CSF. Hence classification is as follows: The hydrocephalus may be due to 1) overproduction of CSF 2) obstructive 3) absorption defect. Depending on the exact aetiology, a secondary classification could be added under the following headings: 1) congenital, 2) acquired, eg; traumatic inflammatory, neoplastic, and degenerative . Bypassing the site of obstruction to CSF flow by diverting the CSF from ventricular cavity to a site where it is readily absorbed is the basic principle underlying the treatment of hydrocephalus. Extensive range of complications has been reported for shunting for hydrocephalus. They could be classified as mechanical or flow-related complications as CSF over drainage leading to subdural hematoma, subdural collections, low-pressure headaches cranial deformity, and asymmetrical drainage can lead to trapping or isolation of a part of a ventricular system. The slit ventricular syndrome is a complication related to absorption. Besides, ascites, loculations, hydrocele, perforation of the stomach, large and small bowel are also described. The success rates of shunt operation for hydrocephalus depend on the age of the patient and the reason why the shunt is needed. Generally, there is around a 50% failure rate for ventriculoperitoneal shunts.

ELIGIBILITY:
Inclusion Criteria:

Patients with borderline hydrocephalus

* Clinically:suspicious and non specific symptoms as

  * Headache
  * Macrocranium
  * Vomiting
  * Gait instability
  * Dementia
  * Urine incontinence.
  * delayed milestone.
* Radiologicaly: dilated ventricular system.

Exclusion Criteria:

* Documented or clinically and radiologically evident cases of hydrocephalus
* Patients known to have contraindications for MRI, e.g. an implanted magnetic device, pacemakers or claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Decompressive changes in CT brain | 2 months
  CT brain showing decompression of the ventricular system in response to ventriculoperitoneal shunt

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Taghyan, Study Chair — professor

REFERENCES:
- [Background] Brassow F, Baumann K. Volume of brain ventricles in man determined by computer tomography. Neuroradiology. 1978;16:187-9. doi: 10.1007/BF00395246. PMID 310977
- [Background] Algin O, Hakyemez B, Parlak M. Phase-contrast MRI and 3D-CISS versus contrast-enhanced MR cisternography on the evaluation of the aqueductal stenosis. Neuroradiology. 2010 Feb;52(2):99-108. doi: 10.1007/s00234-009-0592-x. Epub 2009 Sep 15. PMID 19756563
- [Background] Venkataramana NK. Hydrocephalus Indian scenario - A review. J Pediatr Neurosci. 2011 Oct;6(Suppl 1):S11-22. doi: 10.4103/1817-1745.85704. PMID 22069421
- [Background] Bhatnagar V, George J, Mitra DK, Upadhyaya P. Complications of cerebrospinal fluid shunts. Indian J Pediatr. 1983 Mar-Apr;50(403):133-8. doi: 10.1007/BF02821431. No abstract available. PMID 6618572
- [Background] Reddy GK, Bollam P, Caldito G. Long-term outcomes of ventriculoperitoneal shunt surgery in patients with hydrocephalus. World Neurosurg. 2014 Feb;81(2):404-10. doi: 10.1016/j.wneu.2013.01.096. Epub 2013 Feb 4. PMID 23380280